CLINICAL TRIAL: NCT04338633
Title: Post-operative Pain Reduction After Application of Three Intracanal Medicament Within Necrotic Root Canals and Pulp
Brief Title: Post-operative Pain Reduction
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Minia University (Other)
Responsible Party: Principal Investigator, Mohamed Salah Mohamed Fahmy, PHD Candidate - Endodontic Department- Faculty of Dentistry, Minia University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 314
Record Dates: First submitted 2020-04-06; First posted 2020-04-08 (Actual); Last update posted 2020-04-08 (Actual); Status verified 2020-04

CONDITIONS: Effects of the Elements
MeSH Terms: interventions — UltraCal XS

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Masking Description: double
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Conventional calcium hydroxide paste (Active Comparator): Application of Conventional calcium hydroxide paste
  Interventions: Drug: Conventional calcium hydroxide paste
- Calcium hydroxide nanoparticle (Experimental): Application of Calcium hydroxide nanoparticle
  Interventions: Drug: Calcium hydroxide nanoparticle
- Combined Calcium hydroxide with silver nanoparticle (Experimental): Application of Combined Calcium hydroxide with silver nanoparticle
  Interventions: Drug: Combined Calcium hydroxide with silver nanoparticle

INTERVENTIONS:
Drug: Conventional calcium hydroxide paste — Conventional calcium hydroxide paste (Ultracal) will be removed in second visit.
  Other Names: Ultracal
  Arms: Conventional calcium hydroxide paste
Drug: Calcium hydroxide nanoparticle — Calcium hydroxide nanoparticle. manufactured in NanoTech. institute, will be removed in second visit.
  Arms: Calcium hydroxide nanoparticle
Drug: Combined Calcium hydroxide with silver nanoparticle — Combined Calcium hydroxide with silver nanoparticle will be removed in second visit.
  Arms: Combined Calcium hydroxide with silver nanoparticle

SUMMARY:
Recruited patients with necrotic pulp after application of conventional calcium hydroxide paste are assigned to group, Calcium hydroxide nanoparticle group and Combined Calcium hydroxide with silver nanoparticle group and record postoperative pain afterwards.

DETAILED DESCRIPTION:
The investigator will recruit patients who are found eligible to the criteria, conventional calcium hydroxide paste , Calcium hydroxide nanoparticle and Combined Calcium hydroxide with silver nanoparticle . After 48 hours, patients will be randomly assigned to removal of intracanal medication

After the visit, patients will be asked to record post operative pain by Numerical Rating Scale)in a given sheet

ELIGIBILITY:
Inclusion Criteria:

* • Medically free patients.

  * Patient's age between 25-50 years.
  * Sex includes both male and female.
  * Radiographic evidence of a periapical radiolucent lesion associated with tooth.
  * Necrotic pulp as indicated by thermal pulp testing.
  * No history of previous endodontic treatment of the tooth.

Exclusion Criteria:

* • Teeth with unfavorable conditions for rubber-dam application.

  * Teeth with acute periapical abscesses swelling.
  * Medically compromised patients.
  * Immature teeth with open apices.
  * Multi rooted teeth.
  * Pregnant women.

Ages: 25 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2020-04 (Estimated); Primary Completion 2020-11 (Estimated); Study Completion 2020-11 (Estimated)

PRIMARY OUTCOMES:
change in post operative pain (Visual Analogue Scale) | Intrappointment at 4,24,48,72 and 96 hours ]
  Numerical (0-10)

CONTACTS AND LOCATIONS:
Overall Officials: Magdy Mohamed Aly, Professor, Study Director — Dean of Faculty
Locations (1):
- Faculty of Dentistry, Minia University, Minya, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Singh RD, Khatter R, Bal RK, Bal CS. Intracanal medications versus placebo in reducing postoperative endodontic pain--a double-blind randomized clinical trial. Braz Dent J. 2013;24(1):25-9. doi: 10.1590/0103-6440201302039. PMID 23657409